CLINICAL TRIAL: NCT03874663
Title: Acceptability and Performance of HIV Self-Testing in a Youth Population in Nigeria
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nigerian Institute of Medical Research (Other Government); University of North Carolina, Chapel Hill (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Juliet Iwelunmor, PhD, Professor of Medicine Washington University School of Medicine in St. Louis, Washington University School of Medicine
Other Study IDs: 29882; UG3HD096929 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: HIV Prevention
Keywords: HIV; HIV self-testing; young people; Nigeria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Oral HIV Self-testing: Evaluate the acceptability and performance of a directly assisted oral HIV self-testing (HIVST) in a youth population aged 14-24 in Nigeria
  Interventions: Device: Directly assisted oral HIV self-testing (HIVST)

INTERVENTIONS:
Device: Directly assisted oral HIV self-testing (HIVST) — 1. To determine the ability of participants with unknown HIV status to correctly perform oral HIVST;
  2. To compare the results of the oral HIVST with confirmatory rapid finger prick HIV test.
  3. To explore participants attitudes and preferences towards oral HIVST.
  4. To explore the feasibility, acceptability and appropriateness of using a mobile photo verification app to verify HIV self-testing results.
  Other Names: OraQuick ADVANCE Rapid HIV 1/2 Antibody Test

SUMMARY:
The purpose of this study is to evaluate the acceptability and performance of a directly assisted oral HIV self-testing (HIVST) program in a youth population aged 14-24 in Nigeria. The study is oral HIV self-testing (HIVST) program in a youth population aged 14-24 in Nigeria. The study is focused on assessing young people's ability to correctly perform the test.

DETAILED DESCRIPTION:
Nigerian youth aged 14-24 make up a significant proportion of Sub-Saharan African youth newly diagnosed with HIV. However, they do not access essential HIV prevention services, like routine HIV testing, pre-exposure prophylaxis (PrEP) and sexually transmitted infection (STI) testing.This is partly explained by barriers that are individual (fear, and low perceived risk), social (insufficient social support) and structural (poor access to testing) factors. Additionally, the most affected groups of young people have remained largely unreached by traditional HIV testing services.

HIV self-testing (HIVST) can mitigate some of these barriers by decentralizing HIV testing,decreasing stigma, and linking HIV-negative individuals with preventive services. HIVST is a process in which a person collects his or her own specimen (oral fluid or blood) using a simple rapid HIV test and then performs the test and interprets the result, often in a private setting, either alone or with someone he or she trusts. HIVST offers an alternative to facility-based HIV testing services, particularly for youth populations who may fear to get tested for HIV due to stigma and discrimination. Recognizing the expanding evidence supporting the effectiveness of HIVST, particularly the OraQuick HIV self-testing kits (see Tun et al, 2018; Nagendo et al., 2017; Kurth et al., 2016; Choko et al., 2016; and WHO pre-qualification report under the Publications Tab), the World Health Organization released HIVST guidelines in 2016.

This study is in part with a parent study called ITEST (Innovative Tools to Expand HIV Self-Testing) aimed at developing and implementing innovative youth-friendly HIV self-testing services through open challenges and apprenticeships that provides youth opportunities to learn about social problems (like HIV) that affect their lives and then propose actions to address these problems, informed by the youth participatory action research framework (YPAR).

Recent study conducted in Nigeria, already demonstrate the feasibility and acceptability of HIVST among 257 men sleeping with men (MSMs) in Nigeria (see paper by Tun, 2018). In that study, 97% reported using the HIVST kits. Almost all participants reported that the HIVST kit instructions were easy or somewhat easy to understand (99.6%) and perform the test (98.0%).The most common reasons they liked the test were ease of use (87.3%), confidentiality/privacy (82.1%), convenience (74.1%) and absence of needle pricks (64.9%).

However given the need for youth friendly HIV testing services that are accessible, acceptable, appropriate and effective to address the specialized needs of young people and the public health implications of unknown HIV status, especially among young people, the purpose of this study is to evaluate the acceptability and performance of directly assisted oral HIVST in a youth population in Nigeria.

Given that oral HIV self-testing is a new testing approach in Nigeria, there is a strong need for more research to be done to provide evidence of its acceptability in the general population. Currently, there has been one completed study that assessed the feasibility and acceptability of HIVST; however, this was conducted among a sub-population group (Men who have sex with Men) [Tun et. al., 2018]. Thus, this study seeks to examine in a general population of adolescents and young people, the acceptability and performance of oral HIV self-testing and the factors that influence acceptability.

Study Procedures:

1. Study participants will be recruited from a health facility in Nigeria as well as from local college campuses and other youth-friendly community settings in Nigeria. At the health facilities, study flyers with mobile phone contact numbers will be used to recruit participants along with provider word of mouth. At the schools and college campuses, and community settings, research assistants will introduce the study and participants between the ages of 14-24 will be invited to participate in the study. All participants recruited at the health facility, schools, college campuses, and community settings will be given written informed consent.
2. Following informed consent, study staff will administer a pre-HIV testing questionnaire to collect basic demographic information and assess HIV test history, sexual behavior history, HIV self-testing knowledge, importance, confidence, and concerns with performing the test. Respondents will be given a tablet computer-assisted survey instrument (CASI) due to the sensitive nature of some of questions by NIMR research assistant and are able to enter their responses themselves. This is thought to increase the validity of responses, as respondents are more likely to give truthful answers.
3. Next, instructions on how to perform the oral HIVST using OraQuick Rapid HIV 1⁄2 Antibody, (OraSure Technologies), a rapid oral fluid test kit approved by FDA to detect HIV antibodies, will be given in person to each participant by the research assistant. The research assistant will show a short professionally developed video to introduce the concept of HIVST. The use of the video will allow us to standardize information provided to participants and limit discrepancies in the content and quality of the information provided. Pictorial information on how to perform the test will also be provided to participants. Instructions on how to perform the test will be repeated if asked by participants.
4. Next, participants perform the oral HIVST in the privacy of a separate room or mobile tent-set up. After completion of the test, participants take a photograph of their test results. The photographs of the test result will be taken using a study issued tablet. To login to the tablet, each participant will be provided with a unique login number which corresponds to the ID on their pre and post test. By using the photo verification component, we seek to examine whether they can correctly perform the test on their own and interpret the result, as intended. The trained research assistant will record the results as captured in the photo.
5. Next the trained research assistant from our partner organization, the Nigerian Institute of Medical Research (NIMR), will perform a confirmatory finger prick HIV test according to the national standards using the Determine and Uni-Gold in parallel as per the Nigerian HIV testing country guidelines. In a case where a participant test positive for HIV using the the HIVST kit, confirmatory testing will be available to the participant at the same location immediately.
6. Finally, study participants will complete a post-test questionnaire to capture perceived acceptability of HIVST and whether they had any problems performing oral HIVST. Respondents will complete survey on a tablet computer-assisted survey instrument (CASI) due to the sensitive nature of some of questions by NIMR research assistant and are able to enter their responses themselves.

We will adhere to the WHO five key components-the "5 Cs"-that must be respected and adhered to by all HIV Testing services. These components are: Consent Confidentiality Counselling Correct test results Connection/linkage to prevention, care and treatment.

The five Cs, and the key principles they entail include the following:

1. People being tested for HIV must give informed consent to be tested. They must be informed of the process for HTC, the services that will be available depending on the results, and their right to refuse testing. Mandatory or compulsory (coerced) testing is never appropriate, regardless of where that coercion comes from: health-care providers, partners, family members, employers, or others.
2. Testing services must be confidential, meaning that the content of discussions between the person tested and the health-care worker, testing provider, or counselor, as well as the test results, will not be disclosed to anyone else without the consent of the person tested.
3. Testing services must be accompanied by appropriate and high-quality pre-test information or pre-test counselling, and post-test counselling. Given that the confirmatory testing will be administered immediately at the testing site, our partners NIMR, a PEPFAR supported site will provide pre- and post-test counseling following regulations in Nigeria. NIMR is a PEPFAR Support HIV Care Services in Lagos, Nigeria providing care since 2003 for over 24,000 individuals living with HIV in Lagos, Nigeria.
4. Provision of correct test results. Testing must be performed and quality assurance measures followed according to internationally-recognized testing strategies, norms, and standards based on the type of epidemic. Results must be communicated to the person tested unless that person refuses the results.
5. Connections to HIV prevention, treatment and care and support services should be supported through concrete and well-resourced patient referral, support, and/or tracking systems.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are agree to provide consent
* Residing in Lagos
* Between the ages of 14 to 24 years

Exclusion Criteria:

* Younger than 14 and older than 24
* Inability to comply with study protocol
* Illness, cognitive impairment or threatening behavior with acute risk to self or others
* No informed consent
* Do not reside in Nigeria

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals aged 14-24 years old and residing in Lagos, Nigeria. Individuals who do not know their HIV status because they have never tested or their last HIV test was negative.
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Performance of HIV Self-testing | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 30 minutes for the pre-and-post test HIV questionnaires.
  The ability of participants with unknown HIV status to correctly perform and interpret an oral HIV self-test and compare their results to staff/lab testing.
HIV Self-testing Acceptability | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 30 minutes for the pre-and-post test HIV questionnaires.
  Pre- and post-HIV self-testing importance, confidence, and acceptability

SECONDARY OUTCOMES:
HIV self-testing knowledge | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 30 minutes for the pre-and-post test HIV questionnaires.
  Questions related to HIV self-testing knowledge is included in the pre- and post- questionnaire.
Feasibility of HIV self-testing photo verification app | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 10 minutes to complete the feasibility questions.
  Questions related to the feasibility of whether a photo verification mobile app can be used to verify HIV self-testing results.
Acceptability of HIV self-testing photo verification app | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 10 minutes to complete the acceptability questions.
  Questions related to the acceptability of using a photo verification mobile app to verify HIV self-testing results.
Appropriateness of HIV self-testing photo verification app | Specifically for data collection, we anticipate that the entire study will take 2 hours to complete, 1 hours and 30 minutes for HIV self-testing and confirmatory rapid HIV blood-prick test and 10 minutes to complete the appropriateness questions.
  Questions related to the approproatieness of using a photo verification mobile app to verify HIV self-testing results.

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nigeria Framework. National HIV and AIDS Strategic Framework. 2017-2021.
- [Background] NACA. Federal Republic of Nigeria, Global AIDS Report: Country Progress Report. 2015. Accessed Novembner, 2015.
- [Background] NDHS. National Population Commision; Nigerian Demographic and Health Survey Reports. 2013.
- [Background] Asaolu IO, Gunn JK, Center KE, Koss MP, Iwelunmor JI, Ehiri JE. Predictors of HIV Testing among Youth in Sub-Saharan Africa: A Cross-Sectional Study. PLoS One. 2016 Oct 5;11(10):e0164052. doi: 10.1371/journal.pone.0164052. eCollection 2016. PMID 27706252
- [Background] Sekoni AO, Somefun EO, Fatoba OO, Onajole AT. Use of HIV Screening Services and Sexual Behavior of In-School Adolescents in Surulere LGA, Lagos State. Nig Q J Hosp Med. 2015 Jul-Sep;25(3):202-8. PMID 27295814
- [Background] Sam-Agudu NA, Folayan MO, Ezeanolue EE. Seeking wider access to HIV testing for adolescents in sub-Saharan Africa. Pediatr Res. 2016 Jun;79(6):838-45. doi: 10.1038/pr.2016.28. Epub 2016 Feb 16. PMID 26882367
- [Background] Tucker JD, Wei C, Pendse R, Lo YR. HIV self-testing among key populations: an implementation science approach to evaluating self-testing. J Virus Erad. 2015 Jan;1(1):38-42. doi: 10.1016/S2055-6640(20)31145-6. PMID 26005717
- [Background] Indravudh PP, Sibanda EL, d'Elbee M, Kumwenda MK, Ringwald B, Maringwa G, Simwinga M, Nyirenda LJ, Johnson CC, Hatzold K, Terris-Prestholt F, Taegtmeyer M. 'I will choose when to test, where I want to test': investigating young people's preferences for HIV self-testing in Malawi and Zimbabwe. AIDS. 2017 Jul 1;31 Suppl 3(Suppl 3):S203-S212. doi: 10.1097/QAD.0000000000001516. PMID 28665878
- [Background] Smith P, Wallace M, Bekker LG. Adolescents' experience of a rapid HIV self-testing device in youth-friendly clinic settings in Cape Town South Africa: a cross-sectional community based usability study. J Int AIDS Soc. 2016 Jan;19(1):21111. doi: 10.7448/IAS.19.1.21111. Epub 2016 Dec 23. PMID 28406597
- [Background] Jennings L, Conserve DF, Merrill J, Kajula L, Iwelunmor J, Linnemayr S, Maman S. Perceived Cost Advantages and Disadvantages of Purchasing HIV Self-Testing Kits among Urban Tanzanian Men: An Inductive Content Analysis. J AIDS Clin Res. 2017 Aug;8(8):725. doi: 10.4172/2155-6113.1000725. Epub 2017 Aug 31. PMID 29051841
- [Background] WHO. HIV Testing Services: WHO recommends HIV Self-testing. Geneva2016.
- [Background] Ozer EJ. Youth-Led Participatory Action Research: Developmental and Equity Perspectives. Adv Child Dev Behav. 2016;50:189-207. doi: 10.1016/bs.acdb.2015.11.006. Epub 2016 Jan 25. PMID 26956074
- [Background] Ozer EJ, Piatt AA, Holsen I, Larsen T, Lester J, Ozer EM. INNOVATIVE APPROACHES TO PROMOTING POSITIVE YOUTH DEVELOPMENT IN DIVERSE CONTEXTS. Positive Youth Development in Global Contexts of Social and Economic Change. 2016:12
- [Background] Ozer EJ. Youth-led participatory action research. Handbook of methodological approaches to community-based research: Qualitative, quantitative, and mixed methods. 2016:263-272
- [Background] Cammarota J, Fine M. Revolutionizing education : youth participatory action research in motion. New York, NY: Routledge; 2008
- [Background] Tun W, Vu L, Dirisu O, Sekoni A, Shoyemi E, Njab J, Ogunsola S, Adebajo S. Uptake of HIV self-testing and linkage to treatment among men who have sex with men (MSM) in Nigeria: A pilot programme using key opinion leaders to reach MSM. J Int AIDS Soc. 2018 Jul;21 Suppl 5(Suppl Suppl 5):e25124. doi: 10.1002/jia2.25124. PMID 30033680
- See also: National HIV and AIDS Strategic Framework. 2017-2021 — https://naca.gov.ng/wp-content/uploads/2018/05/National-HIV-and-AIDS-Strategic-Plan-FINAL1.pdf

DOCUMENTS (1):
  • Informed Consent Form (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03874663/ICF_000.pdf